CLINICAL TRIAL: NCT02536885
Title: The Effect of the Perioperative Blood Pressure on the Onset of Postoperative Cognitive Dysfunction in Adults
Brief Title: The Effect of Blood Pressure on the Postoperative Cognitive Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Dostalova Vlasta, MD, PhD, Dostalova Vlasta, MD, PhD, University Hospital Hradec Kralove
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201508-S21P
Record Dates: First submitted 2015-08-27; First posted 2015-09-01 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Mild Cognitive Impairment
Keywords: Postoperative cognitive dysfunction; Blood pressure; Anesthesia
MeSH Terms: conditions — Cognitive Dysfunction; Postoperative Cognitive Complications

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liberal group (Experimental): During the surgery, blood pressure of the patients will be maintained within ± 25% of the patient's normal blood pressure.
  Interventions: Procedure: Liberal group
- Restrictive group (Experimental): During the surgery, blood pressure of the patients will be maintained within ± 10% of the patient's normal blood pressure.
  Interventions: Procedure: Restrictive group

INTERVENTIONS:
Procedure: Liberal group — If the pressure decreases below 75% of patient's baseline mean arterial pressure for more than 1 min, continuous application of noradrenalin will be initiated. If the blood pressure increases above 125% of patient's baseline mean arterial pressure for more than 1 min, Ebrantil (urapidil hydrochlorid) will be applied in dose of 5 mg intravenously with the possibility of repeated doses in 2 minutes intervals.
  Arms: Liberal group
Procedure: Restrictive group — If the pressure decreases below 90% of patient's baseline mean arterial pressure for more than 1 min, continuous application of noradrenalin will be initiated. If the blood pressure increases above 110% of patient's baseline mean arterial pressure for more than 1 min, Ebrantil (urapidil hydrochlorid) will be applied in dose of 5 mg intravenously with the possibility of repeated doses in 2 minutes intervals.
  Arms: Restrictive group

SUMMARY:
Permanent and temporary cognitive impairment in the perioperative period is of great importance to patients. Hypoperfusion due to the intraoperative hypotension is often mentioned as a possible cause of postoperative cognitive dysfunction.

DETAILED DESCRIPTION:
All patients aged above 60 years undergoing planned spinal surgery in the prone position in the duration of 1-3 hours under general anesthesia will be included in the study. In group L (liberal), the value of blood pressure will be corrected with the change of mean arterial pressure (MAP) ± 25% patient's mean arterial pressure, and group R (restrictive) with the change of MAP ± 10%. Cognitive dysfunction tests will be executed on the day before the surgery, two hours after the surgery and on the third postoperative day. Anesthesia will be managed according to the standardised protocol. Concentration of desflurane will be adjusted according to entropy values (target 40-50). Analgetics will be applied according to surgical pleth index (SPI) values. Sufentanil will not be applied in the last 15 minutes. Extubation will be performed at the operating theatre when meeting all extubation criteria including train of four ratio (TOFR) above 92%. Neither syntophyllin, nor pharmacological decurarization (syntostigmin) will be applied to the patients.

ELIGIBILITY:
Inclusion Criteria:

* GCS 15
* ASA risk I - III
* planned spinal surgery in the prone position
* duration of the procedure of 1-3 hours

Exclusion Criteria:

* hypertension above 180/100 torr preoperatively
* blood pressure below 130/80 torr preoperatively

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-09; Primary Completion 2018-06 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Change in cognitive behavior | within the first 3 days after surgery
  measured by Addenbrooks cognitive test

CONTACTS AND LOCATIONS:
Overall Officials: Vlasta Dostalova, MD, PhD, Principal Investigator — University Hospital Hradec Kralove
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Czechia